CLINICAL TRIAL: NCT04231682
Title: A Prospective Randomized Double-Blind, Placebo-Controlled Phase 2 Study Evaluating the Efficacy and Safety of Early Administration of Denosumab 60mg for Prevention and Treatment of Osteoporosis in First-time Liver Transplant Recipients
Brief Title: A Study to Evaluate Efficacy and Safety of Denosumab for Prevention and Treatment of Osteoporosis in 1st Time Liver Transplant Recipients.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Grant support was withdrawn from Amgen Pharmaceuticals
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Catherine Anastasopoulou, MD, PhD, FACE, Attending Physician, Diabetes and Endocrinology., Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-2020-300
Record Dates: First submitted 2020-01-03; First posted 2020-01-18 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Denosumab receiving group. (Experimental): Patients in this arm will receive denosumab injection 60 mg subcutaneously every 6 months. (A total of 4 injections)
  Interventions: Drug: Denosumab Injection
- Placebo receiving group. (Placebo Comparator): Patients in this arm will receive Placebo injection subcutaneously every 6 months. (A total of 4 injections)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Denosumab Injection — Use of denosumab in post liver transplant patient for prevention and management of osteoporosis and bone loss.
  Arms: Denosumab receiving group.
Drug: Placebos — Use of placebo in post liver transplant patient for prevention and management of osteoporosis and bone loss.
  Arms: Placebo receiving group.

SUMMARY:
Organ transplant recipients are known to suffer from bone loss and subsequent fractures after the transplant operation with the most rapid bone loss occurring within the first 3-12 months. Guidelines for prevention and treatment of this serious complication are only written by individual medical societies interested in each organ (separate kidney from liver or heart transplants management) and they are based on studies done with limited medications choices. The majority of studies are done with the use of bisphosphonates, and there are very limited, or no data, on the effect of other medications used for Osteoporosis, including the use of denosumab. This study will focus on the evaluation of the efficacy and safety of denosumab 60mg use early (within first 3 months) after Liver Transplantation in the management of bone loss and prevention of fragility fractures. Different tests will be used to study the effect of the medication on the skeleton, including imaging studies as well as specific labwork.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years old
* First-time Liver transplant Recipients
* All men, postmenopausal women and women with history of hysterectomy or tubal ligation
* Patients who have not been treated with medications for Osteoporosis within the past 12 months before the liver transplant
* Patients able and agreeable to follow up at out Institution for the duration of the study
* Patients hospitalized for less than 45 consecutive days after the liver transplant surgery
* Patients with GFR>30ml/min (calculated by Cockcroft-Gault equation, see Table 3 for details)
* Patients with corrected Calcium >= 8.5
* Patients with PTH intact levels WNL (as per lab values)
* Patients with vit D>=20; NOTE: patients with vit D <20 will be treated with high dose Ergocalciferol 50,000 units daily and rechecked in 2 weeks
* Patients with t-score >=-3.5 at all sites checked by DEXA scan
* Patients agree to sign an informed consent form to be in the study
* Can be treated with denosumab or placebo within 3 months from the liver transplant date

Exclusion Criteria:

* Patients with previous transplants
* Patients that are getting 2 simultaneous transplants, like combined kidney and liver transplants
* Age < 18 year old
* Patients hospitalized for over 45 days after the liver transplant surgery
* Patients with GFR< 30ml/min
* Patients with hypocalcemia defined as corrected calcium < 8.5
* Patients with extensive dental problems, previous hx of Osteonecrosis of the jaw (ONJ) and/or high risk for developing ONJ
* Patients with current Hyperthyroidism
* Patients with current Primary Hyperparathyroidism defined by the combination of elevated calcium and PTH intact levels
* Patients with severe Osteoporosis as defined by t-score <-3.5 at any site shown by DEXA scan
* Women of reproductive age without history of tubal ligation or hysterectomy
* Patients who cannot read or understand the Informed Consent Document or study instructions
* Patients with diagnosis of dementia, or otherwise unable to give informed consent
* Patients unable to follow up in our Institution for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The percentage changes in bone mass calculated by DEXA scan t-score of Lumbar Spine in the intervention and control groups at 12 months. | 12 months

SECONDARY OUTCOMES:
The percentage changes in bone mass calculated by DEXA scan t-score of Femoral Neck, Total Hip and Wrist in the intervention and control groups at 12 months. | 12 months
The percentage changes in bone mass calculated by DEXA scan t-score of Lumbar Spine, Femoral Neck, Total Hip and Wrist in the intervention and control groups at 24 months. | 24 months
The vertebral and non-vertebral fracture incidence at 12 and 24 months. | 12 and 24 months
The percentage changes of biochemical markers of variables of bone turnover (BSAP, CTX and PINP) from baseline to 6, 12, 18 and 24 months after 1st medication administration. | 6, 12, 18 and 24 months
The percentage changes of creatinine, Calcium, Magnesium, Phosphorus, PTH intact and 25-Vit D levels from baseline to 6, 12, 18 and 24 months after the 1st medication administration. | 6, 12, 18 and 24 months
The percentage of patients developing infections, rejection episodes, hospitalizations or ED visits during the study period. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Anastasopoulou, MD, PhD, Principal Investigator — Einstein Medical Center Philadelphia.

IPD SHARING:
Plan to Share IPD: No